CLINICAL TRIAL: NCT01088100
Title: The Correlation Between Certain Clock-gene Genotypes and POCD (Post-operative Cognitive Dysfunction)
Brief Title: Study of the Correlation Between Specific Genes and Cognitive Dysfunction After Surgery
Status: Completed | Type: Observational
Sponsor: Herlev Hospital (Other)
Responsible Party: Melissa Voigt Hansen, Herlev Hospital
Other Study IDs: MVH-01
Record Dates: First submitted 2010-03-12; First posted 2010-03-17 (Estimated); Last update posted 2011-01-10 (Estimated); Status verified 2011-01

CONDITIONS: Genotype; Cognitive Impairment
Keywords: POCD; clock-gene genotypes; HPER3
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Genotype

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Whole blood on filter paper
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with POCD - cases: Out of the 976 patients included in the ISPOCD2 study (Abildstrom H, Christiansen M et al. Apolipoprotein E genotype and cognitive dysfunction after noncardiac surgery. Anesthesiology 2004;101:855-61) the 93 patients with POCD whose blood samples are stored will be included together with 2x93 controls (without POCD), who will be matched by type of surgery, age, education, ASA-score and sex.
  Interventions: Genetic: Genotyping
- Patients without POCD - controls: Out of the 976 patients included in the ISPOCD2 study (Abildstrom H, Christiansen M et al. Apolipoprotein E genotype and cognitive dysfunction after noncardiac surgery. Anesthesiology 2004;101:855-61) the 93 patients with POCD whose blood samples are stored will be included together with 2x93 controls (without POCD), who will be matched by type of surgery, age, education, ASA-score and sex.
  Interventions: Genetic: Genotyping

INTERVENTIONS:
Genetic: Genotyping — Determination of 3 types of clock gene genotypes (HPER 4/4, 5/4, 5/5) on all blood samples

SUMMARY:
The purpose of this study is to determine whether a certain clock-gene (HPER3) with the 5/5 genotype carries a higher risk of post-operative cognitive dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing non-cardiac and non-neurological surgery in either regional or general anesthesia

Exclusion Criteria:

* daily use of major tranquilizers or antipsychotic medication
* known disease of the CNS
* score less than 24/30 points in MMSE

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Out of the 976 patients included in the ISPOCD2 study (Abildstrom H, Christiansen M et al. Apolipoprotein E genotype and cognitive dysfunction after noncardiac surgery. Anesthesiology 2004;101:855-61)100 patients with POCD whose blood samples are stored will be included together with 100 controls (without POCD), who will be matched by type of surgery, age and sex.
Sampling Method: Non-Probability Sample
Enrollment: 279 (Actual)
Dates: Start 2010-08; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
HPER3 genotype | 3 months

SECONDARY OUTCOMES:
Post-operative morbidity | ½ year

CONTACTS AND LOCATIONS:
Overall Officials: Melissa V Hansen, MD, Principal Investigator — Herlev Hospital
Locations (1):
- Herlev Hospital - Gastro unit, Herlev, Denmark

REFERENCES:
- [Background] Abildstrom H, Christiansen M, Siersma VD, Rasmussen LS; ISPOCD2 Investigators. Apolipoprotein E genotype and cognitive dysfunction after noncardiac surgery. Anesthesiology. 2004 Oct;101(4):855-61. doi: 10.1097/00000542-200410000-00009. PMID 15448517
- [Background] Moller JT, Cluitmans P, Rasmussen LS, Houx P, Rasmussen H, Canet J, Rabbitt P, Jolles J, Larsen K, Hanning CD, Langeron O, Johnson T, Lauven PM, Kristensen PA, Biedler A, van Beem H, Fraidakis O, Silverstein JH, Beneken JE, Gravenstein JS. Long-term postoperative cognitive dysfunction in the elderly ISPOCD1 study. ISPOCD investigators. International Study of Post-Operative Cognitive Dysfunction. Lancet. 1998 Mar 21;351(9106):857-61. doi: 10.1016/s0140-6736(97)07382-0. PMID 9525362
- [Derived] Voigt Hansen M, Rasmussen LS, Jespersgaard C, Rosenberg J, Gogenur I. There is no association between the circadian clock gene HPER3 and cognitive dysfunction after noncardiac surgery. Anesth Analg. 2012 Aug;115(2):379-85. doi: 10.1213/ANE.0b013e318253d6b3. Epub 2012 Apr 27. PMID 22543063